CLINICAL TRIAL: NCT05508854
Title: The Effect of Prenatal Genetic Counseling Service on the anxıety Levels of Pregnancy and the Attitudes of Prenatal Diagnostic Tests
Brief Title: The Effect of Prenatal Genetic Counseling Service
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Çiler ÇOKAN DÖNMEZ, Phd, PhD, Mersin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 485
Record Dates: First submitted 2022-08-18; First posted 2022-08-19 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Anxiety; Attitude
Keywords: prenatal genetic counselling; pregnant; anxiety; attitude; nursing
MeSH Terms: conditions — Anxiety Disorders; Behavior

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Prospective, parallel, two arm, randomized controlled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (counselling) group (Experimental): Experimental (counseling) group Prenatal genetic counseling is a consultancy service that covers the evaluation of the risk status of the baby in the mother's womb for diseases, the tests that can be done for the diagnosis of the disease, test results and presentation.A data collection form will be applied to all pregnant women between the ages of 18-49 who applied to the medical genetics polyclinic between September and November 2022 and wished to participate in the study. Prenatal genetic counseling will then be given. When it comes to obtaining genetic results, an individual interview will be made with the pregnant woman and the data collection form will be applied again. In the study, routine clinical information will be given to the pregnant women in the control group by the physician. Before the clinical information and when they come to get genetic results, the data collection form will be applied again by making an individual interview with the pregnant woman.
  Interventions: Genetic: prenatal genetic counselling
- Control group (No Intervention): In the study, routine clinical information will be given to the pregnant women in the control group by the physician. Before the clinical information and when they come to get genetic results, the data collection form will be applied again by making an individual interview with the pregnant woman.

INTERVENTIONS:
Genetic: prenatal genetic counselling — Prenatal genetic counseling is a consultancy service that covers the evaluation of the risk status of the baby in the mother's womb in terms of genetic diseases, the tests and risks that can be done for the diagnosis of the disease, the test results and information about the disease in case of illness and the presentation of options.
  Arms: Experimental (counselling) group

SUMMARY:
The research is planned as a randomized controlled experimental study in order to determine the effect of prenatal genetic counseling service on the anxiety levels and attitudes of pregnant women towards prenatal diagnostic tests and the relationship between these two parameters.

Hypotheses of the Research:

Three different sets of hypotheses were established for the research. First Hypothesis Set; H0: Prenatal genetic counseling service; It has no effect on the anxiety levels experienced by pregnant women.

H1: Prenatal genetic counseling service; have an effect on the anxiety levels experienced by pregnant women.

Second Hypothesis Set; H0: Prenatal genetic counseling service; It has no effect on the attitudes of pregnant women towards screening and diagnostic tests.

H1: Prenatal genetic counseling service; It has an effect on the attitudes of pregnant women towards screening and diagnostic tests.

Third Hypothesis Set; H0: There is no relationship between the anxiety experienced by pregnant women and their attitudes towards screening and diagnostic tests.

H1: There is a relationship between the anxiety experienced by pregnant women and their attitudes towards screening and diagnostic tests.

DETAILED DESCRIPTION:
In the study, it was aimed to determine the relationship between the effect of prenatal genetic counseling service on the anxiety levels of pregnant women and their attitudes towards prenatal diagnostic tests, and the anxiety levels of pregnant women and their attitudes towards prenatal diagnostic tests.

Pregnant women who applied to Adana City Hospital Medical Genetics Outpatient Clinic for prenatal diagnosis and met the research criteria and volunteered to participate in the study will be randomly assigned to the study and control groups according to the block randomization method in order to eliminate the selection bias according to the outpatient clinic list and to ensure the balance in the number of individuals between the groups.

In the study, there will be two groups, the study and the control, selected by randomization. Pregnant women who meet the research criteria will be informed about the research in the Medical Genetics outpatient clinic. Informed (voluntary) consent forms will be signed by the pregnant women who accept to participate in the study.

A data collection form will be applied to all pregnant women participating in the study. Before prenatal genetic counseling is given to the pregnant women in the study group, a data collection form will be applied. Prenatal genetic counseling will then be given. In this consultancy, after giving information about what the diagnostic tests are and their purpose, specific consultancy will be given to the proposed invasive test. When she comes to get genetic results, the data collection form will be applied again by making an individual interview with the pregnant woman. The result of the diagnosis test of the pregnant and the decision to continue or terminate the pregnancy will be recorded in the data collection form. Families who are diagnosed with a disease that threatens the life of the fetus or is incompatible with life will be counseled to receive perinatal palliative care. During this period, they will be guided to communicate with health professionals who can get support and they will be supported to make applications for their spiritual needs. In all these stages, care will be provided to the pregnant with a multidisciplinary approach.

In the study, routine clinical information will be given to the pregnant women in the control group by the physician. Before the clinical information and when they come to get genetic results, the data collection form will be applied again by making an individual interview with the pregnant woman.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the research,

  * Between the ages of 18-49
  * Able to read and write Turkish,
  * Open to communication,
  * First prenatal care at 8-11. taking at the gestational week,
  * Having a singleton pregnancy,
  * Prenatal check-ups will be carried out at the hospital where the research will be conducted,
  * At least primary school graduate,

Exclusion Criteria:

* - Those who do not agree to participate in the research,
* Can't read or write Turkish,
* Unable to communicate
* Pregnant women who continue their antenatal follow-ups in another hospital.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Spielberg State-Trait Anxiety Inventory (STAI I-II) | Data collection form will be applied again before the counseling and when the pregnant woman comes to receive the genetic result (within about 2 weeks).
  The Spielberg state-trait anxiety inventory (STAI I-II) was developed by Spielberg et al. to determine the state and trait anxiety levels of individuals separately. STAI I and II are two separate scales, each consisting of 20 items, with a total of 40 questions. These two scales assess the individual's state and trait anxiety.
  The total score obtained from each scale can vary between 20 and 80. A large score indicates a high level of anxiety and a small score indicates a low level of anxiety. The Cronbach's alpha value was found to be between 0.83 and 0.87 for the state anxiety scale, and between 0.94 and 0.96 for the trait anxiety scale.
Prenatal Screening and Diagnostic Test Attitude Assessment Scale | Data collection form will be applied again before the counseling and when the pregnant woman comes to receive the genetic result (within about 2 weeks).
  It is a 4-question scale created by Martetau et al. to evaluate the thoughts of pregnant women about their participation in prenatal diagnosis and screening tests. In the original of the scale, the statements were evaluated over 7 points. It is a good idea (7 points), bad idea (1 point); useful (7 points), not useful (1 point); harmful (1 point), not harmful (7 points); a bad idea (1 point), not a bad idea (7 points) were asked to rate between 1 and 7 points. One point represents a negative attitude, while 7 points represents a highly positive attitude. . The highest score to be obtained from this scale is 28, and the lowest score is 4. The cronbach alpha value of the original scale was found to be 0.83.

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Sarıcam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yesilcinar I, Seven M, Pasalak SI, Guvenc G. Interventions aiming to improve informed decision on prenatal screening and testing: A scoping review of the literature. J Genet Couns. 2021 Dec;30(6):1512-1521. doi: 10.1002/jgc4.1437. Epub 2021 Jun 17. PMID 34137487